CLINICAL TRIAL: NCT05948566
Title: Strategy for Improving Stroke Treatment Response (SISTER) Trial
Brief Title: Strategy for Improving Stroke Treatment Response
Acronym: SISTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Sciences, Inc. (Industry)
Collaborators: University of Cincinnati (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medical University of South Carolina (Other); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS23-U202; UH3NS125023 (NIH)
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Model Description: The first 50 subjects will be randomized equally to the five arms. Response Adaptive Randomization updates will occur every 50 subjects, thereafter, (favoring doses with maximum utility). For each block of 50 subjects, 13 will be allocated to control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: TS23
- Dose 1 TS23 (Experimental): low dose
  Interventions: Biological: TS23
- Dose 2 TS23 (Experimental): next higher dose
  Interventions: Biological: TS23
- Dose 3 TS23 (Experimental): next higher dose
  Interventions: Biological: TS23
- Dose 4 TS23 (Experimental): highest dose
  Interventions: Biological: TS23

INTERVENTIONS:
Biological: TS23 — Monoclonal antibody

SUMMARY:
SISTER is a Phase-II, prospective, randomized, placebo-controlled, blinded, dose finding trial that aims to determine the safety and preliminary efficacy of TS23, a monoclonal antibody against the alpha-2 antiplasmin (a2-AP), in acute ischemic stroke.

DETAILED DESCRIPTION:
SISTER is a Phase II, Bayesian, adaptive, randomized, dose-finding trial of TS23 in patients with acute ischemic stroke. Patients with an anterior cerebral circulation acute ischemic stroke and present between 4.5 to 24 hours of their last known well with a presenting NIH Stroke Scale Score >/=4 (with the patient having a clearly disabling deficit if the NIHSS is 4 or 5) and an imaging evidence of salvageable brain tissue will be eligible and will be approached for an informed consent for study participation. After informed consent is provided, the study will randomize to 4 doses of TS23 and placebo. The trial will enroll up to 300 subjects at up to 60 participating US sites and up to 17 Canadian sites.

The effects of TS23 will be evaluated on two following primary outcomes using a utility function: 1) primary safety outcome: any intracerebral hemorrhage at 30 (+/-4) hours and 2) primary efficacy outcome: NIH Stroke Scale score at 30 (+/-4) hours after drug administration. The study will follow participants for 90 (+/-7) days.

Primary Objective: To identify a dose of TS23 that is safe and more efficacious than placebo for the treatment of patients from 4.5 to 24 hours of last known well, who have evidence of core-penumbra mismatch on perfusion imaging and are not a candidate for standard of care reperfusion therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Suspected anterior circulation acute ischemic stroke
3. NIH Stroke Scale score ≥4 prior to randomization

   a. The participant must have a clearly disabling deficit if NIHSS is 4-5.
4. Favorable baseline neuroimaging consisting of all of the following:

   1. ASPECTS of 6 or more on CT (or ASPECTS of ≥7 on MRI)
   2. Favorable perfusion imaging on CT perfusion (CTP)/MR-perfusion weighted imaging (PWI) consisting of all of the following:

   i. Mismatch ratio of penumbra: core >1.2 ii. Mismatch volume >10 cc iii. Core <70 cc

   c. If CT hypodensity is present, then in the investigator's visual assessment, the total acute infarct volume combined area of (a) the CT hypodensity and (b) the perfusion-based core volume (CBF<30%) should be smaller than perfusion-based volume (area of Tmax>6s minus CBF<30%).
5. Able to receive assigned study drug within 4.5 to 24 hours of stroke onset or last known well.
6. Able to receive assigned study drug within 120 minutes of qualifying perfusion imaging. *
7. Informed consent for the study participation obtained from participant or their legally authorized representatives.

   * Study drug administration is encouraged within 90 minutes after qualifying perfusion image but is allowed up to 120 minutes. After 120 minutes, another perfusion image to ensure that inclusion criteria are met is required.

Exclusion Criteria:

1. Received endovascular treatment with clot engagement.

   1. Patients who undergo groin puncture but clot engagement is not attempted due to spontaneous distal migration are permitted to be enrolled in the trial if all other eligibility criteria are met.
   2. Patients who undergo groin puncture but clot is not engaged due to reasons other than spontaneous distal migration are NOT permitted.
2. Received or planned to receive intravenous thrombolysis.
3. Pre-stroke modified Rankin score >2.
4. Previous treatment with TS23 or known previous allergy to antibody therapy.
5. Known pregnancy, women who are breastfeeding or plan to breastfeed within 3 months of receiving TS23 or have a positive urine or serum pregnancy test for women of childbearing potential.
6. Known previous stroke in the past 90 days.
7. Known previous intracranial hemorrhage, intracranial neoplasm, subarachnoid hemorrhage, or arterial venous malformation.
8. Known active diagnosis of intracranial neoplasm.
9. Clinical presentation suggestive of a subarachnoid hemorrhage, even if initial CT scan was normal.
10. Surgery or biopsy of parenchymal organ in the past 30 days.
11. Known trauma with internal injuries or persistent ulcerative wounds in the past 30 days.
12. Severe head trauma in the past 90 days.
13. Persistent systolic blood pressure >180mmHg or diastolic blood pressure >105mmHg despite best medical management.
14. Serious systemic hemorrhage in the past 30 days.
15. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with International Normalized Ratio (INR) >1.7.
16. Platelets <100,000/mm3.
17. Hematocrit <25 %.
18. Elevated aPTT above laboratory upper limit of normal.
19. Creatinine > 4 mg/dl, or patients receiving renal dialysis, regardless of creatinine.
20. Received the following within the previous 24 hours:

    1. If patient received unfractionated heparin within the last 24 hours, the patient must have an aPTT within normal range prior to enrollment.
    2. Low molecular weight heparins such as Dalteparin, enoxaparin, tinzaparin in full dose within the previous 24 hours.
21. Received Factor Xa inhibitors (such as Fondaparinux, apixaban or rivaroxaban) within the past 48 hours.
22. Received direct thrombin inhibitors (e.g., argatroban, dabigatran, bivalirudin, desirudin, lepirudin) within 48 hours.
23. Received glycoprotein IIb/IIIa inhibitors within the past 14 days.
24. Known pre-existing neurological or psychiatric disease which would confound the neurological/functional evaluations.
25. Current participation in another research drug treatment protocol (i.e., participants could not start another experimental agent until after 90 days).
26. Concurrent acute myocardial infarction, pulmonary embolism, deep venous thrombosis or other thrombotic event that requires anticoagulation or anti-platelet treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with ANY intracerebral hemorrhage (ICH) | At 30 (+/- 4) hours after study drug
  Any ICH visualized on the follow-up CT scan
Stroke severity as measured by the National Institutes of Health Stroke Scale (NIHSS) | At 30 (+/- 4) hours after study drug
  NIHSS is a stroke severity score that ranges from 0 to 42, with higher numbers indicating a more severe stroke. The NIHSS will be adjusted for the baseline value in analysis.

SECONDARY OUTCOMES:
Improvement in level of global disability measured by modified Rankin Score (mRS distribution) | 90 (±7) days
  The modified Rankin Score assessment is a 7-level disability scale that measures the degree of disability or dependence in daily activities of people who have suffered a stroke. Range 0= no disability and 6=dead.
Frequency of Modified Rankin (mRS) score of 0-1 or returning to pre-stroke mRS. | Proportion of patients with modified Rankin scale score 0-1 or return to pre-stroke mRS at 90 (+/-7) days.
  Proportion of patients with modified Rankin scale score 0-1 or return to pre-stroke mRS.
NIHSS | 72 (±12) hours (or at discharge if sooner) after study drug administration.
  NIHSS is a stroke severity score that ranges from 0 to 42, with higher numbers indicating a more severe stroke. The NIHSS will be adjusted for the baseline value in analysis.
α2-antiplasmin (a2AP) level in plasma | at 3 (±1) h after completion of study drug administration
  A serine protease inhibitor responsible for inactivating plasmin.
Matrix metalloproteinase-9 level in plasma | 3 (±1) h after completion of study drug
  An enzyme that regulates the pathological remodeling process that involve inflammation and fibrosis associated with cardiovascular disease.
% brain tissue reperfusion | 30 (±4) h after study drug administration
  Proportion of brain tissue that is reperfused on the follow-up perfusion scan compared to the baseline, calculated as:
  ([baseline minus follow up perfusion imaging area of hypoperfusion]/ baseline area of hypoperfusion); hypoperfusion=T max>6 seconds
Pharmacokinetic analyses | 3 (±1) h, 30 (±4) h, 30 (±5) days & 90 (±7) days after study drug administration. At 90 (±7) days for approximately 50 mITT participants. After approximately 50 mITT participants, it will be obtained at 72h(+12 hrs)/discharge visit, whichever comes 1st.
  Measure of plasma concentrations of TS23
Evaluation of anti-drug antibodies | will be measured at baseline and 90 (±7) days follow-up visit for approximately 50 mITT participants.
  commonly used for characterization of therapeutic antibodies
Proportion of patients with symptomatic intracerebral hemorrhage | 30 (±4) h of study drug administration
  a blood clot large enough to cause significant neurological deterioration.
Proportion of patients with non-intracerebral hemorrhage major or clinically relevant non-major bleeding | 30 days of study drug administration.
  major and non-major events of bleeding that is not in the brain
Plasma fibrinogen level | 3 (±1) h after completion of study drug
  Clotting factor
Proportion of patients with non-bleeding severe adverse events | 90 (±7) days
  Assessment of untoward events
Proportion of patients with stroke-related and all-cause deaths | 90 (±7) days
  measure of important patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Eva Mistry, MBBS, Principal Investigator — University of Cincinnati
Locations (52):
- United States (52):
  - University of Alabama Hospital, Birmingham, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - UCSD Health La Jolla, La Jolla, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Sutter Medical Center, Sacramento, California
  - UCSD Medical Center- Hillcrest Hospital, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - UF Health Shands Hospital, Gainesville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Baptist Healthcare System, Inc., Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - M Health Fairview Ridges Hospital, Burnsville, Minnesota
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - JFK Medical Center, Edison, New Jersey
  - NYU Langone Health, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai West, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Saint Luke's Hospital of Bethlehem Pennsylvania, Bethlehem, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Prisma Health Greenville Memorial, Greenville, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - UVA Medical Center, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Ascension Columbia St. Mary's Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The SISTER trial will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research, and the StrokeNet SOP (ADM 03) regarding results publication. Manuscripts and abstracts that use data from SISTER require approval from the Publication Committee of an original proposal before the concept may proceed. All publications will include this acknowledgement: "Research reported in this publication was supported by the National Institute of Neurological Disorders and Stroke of the National Institutes of Health under Award Number [to be determined]. The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institutes of Health."